CLINICAL TRIAL: NCT03673007
Title: Michigan Contraceptive Access, Research, and Evaluation Study
Brief Title: Michigan Contraceptive Access, Research, and Evaluation Study: Phase 1
Acronym: M-CARES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Opinion Research Center (Other)
Responsible Party: Principal Investigator, Martha Bailey, Adjunct Research Professor, Population Studies Center, Institute of Social Research, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M-CARES
Record Dates: First submitted 2018-08-15; First posted 2018-09-17 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy
Keywords: contraception; financial access to reproductive health care; unintended pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental): Women in this arm of the study receive a voucher which can be used to buy contraception and related services at Planned Parenthood
  Interventions: Behavioral: Gift card to be used for contraceptives that is valued at 50% of cost of name-brand IUD (August 26, 2018-March 3, 2019); Behavioral: Gift card to be used for contraceptives that is valued at 100% of cost of name-brand IUD (March 4, 2019-March 31, 2023)
- Control Group (No Intervention): Women in this arm of the study DO NOT receive a voucher for contraceptives. Women in this arm receive the Planned Parenthood standard of care priced according to the Planned Parenthood sliding scale.

INTERVENTIONS:
Behavioral: Gift card to be used for contraceptives that is valued at 50% of cost of name-brand IUD (August 26, 2018-March 3, 2019) — M-CARES will randomize allocation of vouchers (gift cards) for contraception valued up to 50% of inserting a name-brand IUD (e.g., Skyla, Paraguard, Mirena) for women with out of pocket costs at Planned Parenthood. This intervention occurred between August 18, 2018, and March 3, 2019.
  Arms: Treatment Group
Behavioral: Gift card to be used for contraceptives that is valued at 100% of cost of name-brand IUD (March 4, 2019-March 31, 2023) — M-CARES will randomize allocation of vouchers (gift cards) for contraception valued up to 100% of inserting a name-brand IUD (e.g., Skyla, Paraguard, Mirena) for women with out of pocket costs at Planned Parenthood. This intervention occurred after March 3, 2019.
  Arms: Treatment Group

SUMMARY:
M-CARES will use large-scale administrative data complemented by follow-up surveys and a randomized control trial (RCT) to estimate the causal impact of greater financial access to contraception on a comprehensive set of outcomes. Outcomes include contraceptive use, pregnancy, childbearing, and parenting strategies; partnership decisions and relationship quality; health and health care use; education, labor market success, and public assistance receipt; financial security; neighborhood quality; mental health and stress; and life plans. The resulting estimates will inform a more complete understanding of the costs and benefits of financial access to contraception and, therefore, the investment value of related policies and programs.

ELIGIBILITY:
Inclusion Criteria:

M-CARES will recruit 5,000 women at Michigan Planned Parenthood of Michigan (PPMI) clinics who face potentially large out-of-pocket costs for highly effective contraceptives, especially LARC methods. In order to be eligible to participate in the study, the woman needs to meet the following criteria:

1. . 18-35 years old,
2. . physically capable (biologically female and fecund) and at risk of having a pregnancy (has sex with men),
3. . not pregnant at the time of enrollment and not wishing to become pregnant in the next 12 months,
4. . face some out-of-pocket costs for contraceptives at PPMI

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4633 (Actual)
Dates: Start 2018-08-26 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of patients billing for use of any contraception (1 for use of contraception/0 no use of contraception) | 100 days from enrollment
  Share of participants that purchase contraception as determined by Planned Parenthood of Michigan (PPMI) billing records and code the outcome based on purchases of contraceptives within 100 days of study enrollment (0 for no use of contraception; 1 for use of contraception).
Incidence of patients billing for long-run acting, reversible contraception (LARC) (0 no use of LARC/1 for use of LARC) | 100 days from enrollment
  Share of participants that purchase long-run, acting reversible contraception as determined by PPMI billing records and code the outcome based on purchases of for long-run acting, reversible contraception (LARC) within 100 days of enrollment (0 for no use of contraception; 1 for use of contraception)
Incidence of patients billing for long-run acting, reversible contraception (LARC) (0 no use of LARC/1 for use of LARC) | Up to 1 year post enrollment
  Share of participants that purchase long-run, acting reversible contraception as determined by PPMI billing records and code the outcome based on purchases of for long-run acting, reversible contraception (LARC) up to 1 year of enrollment (0 for no use of contraception; 1 for use of contraception)
Incidence of pregnancy up to 1 year post enrollment | Up to 1 year post-enrollment
  Incidence of pregnancies within one year of enrollment in the study. This data is obtained from PPMI records for pregnancy tests, emergency contraception, abortion, and childbirth as well as surveys.
Incidence of pregnancy up to 3 years post enrollment | Up to 3 year post-enrollment
  Incidence of pregnancies within 3 years of enrollment in the study. This data is obtained from PPMI records for pregnancy tests, emergency contraception, abortion, and childbirth as well as surveys.
Incidence of childbirth up to 1 year post enrollment | Up to 1 years post enrollment
  Incidence of childbirth up to 1 year after enrollment in the study. This data is obtained from PPMI records childbirth and prenatal care, state of Michigan records on natality, and surveys of participants.
Incidence of childbirth up to 3 year post enrollment | Up to 3 years post enrollment
  Incidence of childbirth up to 3 year after enrollment in the study. This data is obtained from PPMI records childbirth and prenatal care, state of Michigan records on natality, and surveys of participants.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Planned Parenthood - Ann Arbor-West, Ann Arbor, Michigan
  - Planned Parenthood - Detroit, Detroit, Michigan
  - Planned Parenthood - Ferndale, Ferndale, Michigan
  - Planned Parenthood - Grand Rapids, Grand Rapids, Michigan
  - Planned Parenthood - Kalamazoo, Kalamazoo, Michigan
  - Planned Parenthood - Lansing, Lansing, Michigan
  - Planned Parenthood - Livonia, Livonia, Michigan
  - Planned Parenthood - Traverse City, Traverse City, Michigan
  - Planned Parenthood - Warren, Warren, Michigan

IPD SHARING:
Plan to Share IPD: No